CLINICAL TRIAL: NCT01398605
Title: Physical Activity and Exercise Dose-response on Cardiovascular Risk Factors in Postmenopausal Women
Brief Title: Physical Activity in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Ying-Tai Wu, School and Graduate Institute of Physical Therapy, College of Medicine, National Taiwan University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 200709026R
Record Dates: First submitted 2011-07-14; First posted 2011-07-20 (Estimated); Last update posted 2011-08-18 (Estimated); Status verified 2011-07

CONDITIONS: Postmenopausal Disorder
Keywords: Postmenopausal women; Physical activity; Cardiovascular risks; Cardiac function; Dose-response
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- moderate exercise training (Experimental)
  Interventions: Other: Exercise training
- intensive exercise training (Experimental)
  Interventions: Other: Exercise training
- Control (No Intervention)

INTERVENTIONS:
Other: Exercise training — Different dose of exercise training
  Arms: intensive exercise training; moderate exercise training

SUMMARY:
The study is designed to investigate the physical activity and its dose-response relationship in postmenopausal women on the cardiovascular risks and cardiac function.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women aged 40 to 80 years and age matched men without major diseases

Exclusion Criteria:

* Known cardiac disease, excessive weight change during last year, cancer and mental disorders

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Body mass index (BMI) | 3 months
Waist circumference | 3 months
Lab data (lipid profile, CRP, insulin resistance) | 3 months
QT interval and corrected QT interval (QTc) | 3 months
Cardiovascular fitness | 3 months
Heart rate recovery after exercise test | 3 months

SECONDARY OUTCOMES:
Myocardial perfusion

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Tai Wu, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan